CLINICAL TRIAL: NCT05950074
Title: Update and Digitalization of a Universal School-based Prevention Intervention for Drug Initiation and Use: the "It´s Up To You" Program
Brief Title: It´s Up To You: Update and Digitalization of a Universal School-based Prevention Intervention for Drug Initiation and Use
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Europeo de Estudios en Prevención (Other)
Collaborators: University of Santiago de Compostela (Other); University of Oviedo (Other); University of the Balearic Islands (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021F055 Tu decides
Record Dates: First submitted 2023-06-20; First posted 2023-07-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Substance Use; Behavior, Addictive; Smoking Behaviors; Alcohol Drinking; Illicit Drug Use
MeSH Terms: conditions — Substance-Related Disorders; Behavior, Addictive; Smoking; Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "It´s Up To You" program (Experimental): Participants will receive the prevention program "It´s Up To You" during the academic year in school hours.
  Interventions: Behavioral: "It´s Up To You" program
- Control (No Intervention): The control group will receive the usual teaching activities regarding substance use prevention.

INTERVENTIONS:
Behavioral: "It´s Up To You" program — The main goal of this program is to prevent substance use and engagement in addictive behaviors through enabling teenagers to make informed and responsible decisions. It seeks to support students in the anticipation of realistic choice situations and problems typically affecting this age group. It is based on social influences, considering the peer group influences (peer pressure) and the affective and cognitive factors that intervene at the time of decision-making and problem-resolution. This program is intended to be delivered by trained teachers in six sessions through six different modules.
  Arms: "It´s Up To You" program

SUMMARY:
This non-randomized cluster-controlled trial examines the effectiveness of the digitalized and updated version of the It´s Up To You - program, a universal school-based prevention intervention for drug initiation and use targeting youth aged between 12 and 17 years.

DETAILED DESCRIPTION:
The goal of this non-randomized cluster-controlled trial targeting youth aged between 12 and 17 years is to examine whether the updated and digitalized version of the preventive intervention named "It´s Up To You" program is effective in preventing drug use initiation and reducing drug use.

Participants in the experimental group will receive 6 sessions conducted by trained teachers. Each session will target a program module about the following topics: (1) What about drugs? (2) A way to start (3) Ana has fun (4) What do you connect to (about the use of the internet and social networks)? (5) Two versions of the same story, and (6) How do my parents come in?

Researchers will compare the experimental group receiving the "It´s Up To You" program to a control group receiving the usual teaching activities regarding substance use prevention. The main goal is to see if participants in the experimental group report lower substance (alcohol, tobacco, and cannabis) use and initiation after the intervention and at a 3-month follow-up related to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Schools having secondary education
* Schools located in Spain.
* Schools willing to participate under the conditions of the study

Exclusion Criteria:

* Schools applying the original "It´s Up To You" prevention program

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Substance use: Alcohol | Past 30-day period
  Items from the survey on drug use in secondary education in Spain for the National Plan on Drugs
Substance use: Tobacco | Past 30-day period
  Items from the survey on drug use in secondary education in Spain for the National Plan on Drugs
Substance use: Cannabis | Past 30-day period
  Items from the survey on drug use in secondary education in Spain for the National Plan on Drugs

SECONDARY OUTCOMES:
Attitudes toward substance use | Past 30-day period
  Attitudes towards drug use Scale
Intention to use alcohol | Next 30-day period
  Intention to drug use in the next month Scale
Intention to use tobacco | Next 30-day period
  Intention to drug use in the next month Scale
Intention to use cannabis | Next 30-day period
  Intention to drug use in the next month Scale
Academic performance | Past 12-months period
  Assessed as having repeated grades
Emotion regulation | Past 30-day period
  Cognitive Emotion Regulation Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Montserrat Juan, PhD, Principal Investigator — Instituto Europeo de Estudios en Prevención
Locations (1):
- Instituto Europeo de Estudios en Prevención, Palma de Mallorca, Spain

REFERENCES:
- [Derived] Castano Y, Gervilla E, Martinez-Vispo C, Juan M, Garcia-Pazo P, Al-Halabi S, Becona E, Calafat A. Effectiveness of a School-Based Drug Prevention Program: Tu Decides 2.0. J Prev (2022). 2025 Nov 17. doi: 10.1007/s10935-025-00883-6. Online ahead of print. PMID 41247593